CLINICAL TRIAL: NCT02459054
Title: SynCardia 50cc Temporary Total Artificial Heart (TAH-t) as a Bridge to Transplant
Brief Title: Syncardia 50cc TAH-t as a Bridge to Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 50cc TAH-t received FDA approval March 5, 2020.
Sponsor: SynCardia Systems. LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-551
Record Dates: First submitted 2014-12-04; First posted 2015-06-01 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure, Right-Sided; Cardiac Failure; Heart Failure, Left-Sided
Keywords: Artificial Heart; Biventricular Heart Failure; SynCardia
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Primary Pediatric Arm (Experimental): Cardiac transplant-eligible pediatric patients at imminent risk of death from biventricular failure who are 10 - 18 years old at time of TAH-t implant. The intervention is implantation with the 50cc temporary Total Artificial Heart as a bridge to transplantation.
  Interventions: Device: SynCardia 50cc temporary Total Artificial Heart (TAH-t)
- Primary Adult Arm (Experimental): Cardiac transplant-eligible adult patients at imminent risk of death from biventricular failure who are 19 - 75 years old at time of TAH-t implant. The intervention is implantation with the 50cc temporary Total Artificial Heart as a bridge to transplantation.
  Interventions: Device: SynCardia 50cc temporary Total Artificial Heart (TAH-t)
- Secondary Arm (Experimental): Cardiac transplant-eligible pediatric and adult patients at imminent risk of death from biventricular failure who do not meet enrollment criteria for a Primary Arm, but meet less restrictive enrollment criteria for the Secondary Arm. The intervention is implantation with the 50cc temporary Total Artificial Heart as a bridge to transplantation.
  Interventions: Device: SynCardia 50cc temporary Total Artificial Heart (TAH-t)

INTERVENTIONS:
Device: SynCardia 50cc temporary Total Artificial Heart (TAH-t) — Replacement of both ventricles and all four valves with the investigational device as a bridge to transplantation.

SUMMARY:
The primary objective of the study is to evaluate whether the 50cc TAH-t can safely support, and provide probable benefit to, transplant-eligible pediatric patients (aged 10 - 18 years) and can safely and effectively support transplant-eligible adult patients (aged 19 - 75 years) at imminent risk of death from biventricular failure without experiencing permanent disabling, stroke-related deficits.

The study will be conducted as a three-arm trial of the 50cc temporary Total Artificial Heart (TAH-t) as a bridge to transplant:

* The Primary Pediatric Arm of the trial will evaluate the safety and probable benefit of the 50cc TAH-t for transplant-eligible patients 10 through 18 years of age.
* The Primary Adult Arm of the trial will evaluate the safety and efficacy of the 50cc TAH-t for transplant-eligible patients 19 through 75 years of age.
* The Secondary Arm will capture pediatric and adult subjects who did not meet enrollment criteria for a Primary Arm, but meet the less restrictive Secondary Arm enrollment criteria, in order to further characterize the use of the device.

DETAILED DESCRIPTION:
Heart failure is the reduced ability of the native heart to pump blood and maintain normal bodily function. Heart transplantation is the standard of care treatment for end-stage heart failure but the supply of donor hearts is insufficient to meet the need and many patients are not eligible for transplantation because of age or comorbid conditions.

On 15 October 2004, the SynCardia 70cc temporary TAH-t System received Food and Drug Administration (FDA) approval for Premarket Approval Application (PMA) #P030011 for in-hospital use as a bridge to transplant (BTT) in cardiac transplant-eligible candidates at risk of imminent death from biventricular failure. The system consists of the implantable TAH-t and an external pneumatic driver. Subsequent to the original approval, two additional external pneumatic drivers have been approved for use with the 70cc TAH-t.

On 30 January 2013, FDA granted a Humanitarian Use Designation (HUD) to the 50cc TAH-t for use as BTT in pediatric patients with biventricular heart failure who have a body surface area (BSA) that can sufficiently accommodate the device. To evaluate the ability of the device to support patients who are too small to be supported with the 70cc TAH-t, SynCardia will conduct a clinical study.

The study will be conducted as a three-arm trial of the 50cc temporary Total Artificial Heart (TAH-t) as a bridge to transplant:

* The Primary Pediatric Arm of the trial will evaluate the safety and probable benefit of the 50cc TAH-t for transplant-eligible patients 10 through 18 years of age.
* The Primary Adult Arm of the trial will evaluate the safety and efficacy of the 50cc TAH-t for transplant-eligible patients 19 through 75 years of age.
* The Secondary Arm will capture pediatric and adult subjects who did not meet enrollment criteria for the pediatric arm, but meet the less restrictive Secondary Arm enrollment criteria, in order to further characterize the use of the device.

Pediatric subject data through six months post-implant will be reported to FDA to support a Humanitarian Device Exemption (HDE) application for an orphan indication in pediatric patients for which there is no alternative replacement device. Pediatric subjects (enrolled in the Primary Pediatric Arm or Secondary Arm) who are continuing on TAH-t support at the six month study visit will continue to be followed under the study every six months until transplant, withdrawal from the study, all subjects in the respective arm have reached an endpoint, or death, whichever occurs first.

The primary objective of the Primary Pediatric Arm of the study is to evaluate whether the 50cc TAH-t can safely support, and provide probable benefit to, transplant-eligible pediatric patients at imminent risk of death from biventricular failure without experiencing permanent disabling, stroke-related deficits. Probable benefit will be measured as transplanted during the first six months, or survival at six months and continuing on support on the initially placed 50cc TAH-t, without experiencing permanent disabling stroke-related deficits.

Safety will be evaluated by the characterization of the adverse event (AE) profile through the six month study end date. AEs will be identified by the terms and definitions of the Pedimacs/Intermacs Registry. The secondary endpoints to establish safety for both the pediatric and adult arms will be measured by performance goals (based on prior experience with the 70cc TAH-t) for the four adverse event categories that are likely to delay or preclude transplant. The four categories are: Major infection (sepsis), Neurological event (CVA), Chronic renal dysfunction, Major device failures/malfunctions per the Pedimacs/Intermacs AE definitions.

Adult patient data through six months post-implant will be reported to FDA to support a Premarket application (PMA) for treatment of small-statured adult patients who are unable to accommodate the 70cc TAH-t in their chest cavity and for whom there is no alternative replacement device. Adult subjects (enrolled in the Primary Adult Arm or the Secondary Arm) will be followed through six months post-implant and, if continuing on support at that time, will continue to be followed under the study every six months until transplant, withdrawal from the study, all subjects in the respective arm have reached an endpoint, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria (Primary Pediatric and Adult Arms):

* At imminent risk of death from biventricular heart failure
* Aged 10 - 18 years (pediatric); 19 - 75 years (adults) at time of implant
* With two functional atrioventricular (A-V) valves
* With Body Surface Area (BSA) of 1.2 through 1.85m2
* With adequate sternum to T10 distance OR Adequate room in chest as determined by 3-D imaging assessment or by other standard clinical assessments

Exclusion Criteria:

* Patients who are not cardiac transplant-eligible
* Cardiac transplant-eligible patients

  * Who cannot be adequately anticoagulated on the TAH-t
  * With insufficient space in the chest
  * Who are on extracorporeal membrane oxygenation (ECMO) support > 3 days
* Patients who are being supported by an investigational device at the time of evaluation for a 50cc TAH-t
* Patients who have required cardiopulmonary resuscitation (CPR) for > 30 minutes within 14 days prior to proposed implant
* Patients who have experienced a stroke within 30 days prior to proposed implant
* Patients who are dialysis-dependent at time of proposed implant

Inclusion Criteria, Secondary Arm (pediatric and adult patients)

* Not eligible for Primary Arm
* At imminent risk of death from biventricular heart failure
* With Body Surface Area (BSA) of 1.2 through 1.85m2
* With adequate sternum to T10 distance OR Adequate room in chest as determined by 3-D imaging assessment or by other standard clinical assessments

Exclusion Criteria, Secondary Arm:

* Patients who are not cardiac transplant-eligible
* Cardiac transplant-eligible patients

  * Who cannot be adequately anticoagulated on the TAH-t
  * With insufficient space in the chest
* Patients who are being supported by an investigational device at the time of evaluation for a 50cc TAH-t

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Probable Benefit (for Pediatric Arm); Efficacy (for Adult Arm) | 6 months
  Probable benefit will be measured at six months post-implant as either transplanted during the first six months, or continuing on support at six months on the same 50cc TAH-t, without experiencing permanent disabling stroke-related deficits.

SECONDARY OUTCOMES:
Safety: Performance Goal of Four Adverse Event Categories | Six months
  Safety will be measured by comparison of rate of occurrence of Major infection (sepsis), Neurological event (CVA), Chronic renal dysfunction, and Major device failures/malfunctions against individual performance goals (based on prior 70cc TAH-t experience).

CONTACTS AND LOCATIONS:
Overall Officials: David Morales, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Francisco Arabia, MD, Principal Investigator — Cardiac-Dynamics
Locations (26):
- United States (26):
  - Banner University Medical Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Indiana University Health, Indianapolis, Indiana
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Strong Memorial Hospital - Paul Yu Heart Center, Rochester, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - The Milton S Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Children's Health of Dallas, Dallas, Texas
  - Baylor University Medical Center at Dallas, Dallas, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Methodist DeBakey Heart and Vascular Center, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Aurora St. Luke's Hospital, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin